CLINICAL TRIAL: NCT00005340
Title: Hypertension in Blacks of West African Origin
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4202; R01HL045508 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity

SUMMARY:
To continue an international collaborative study on hypertension in populations of West African origin.

DETAILED DESCRIPTION:
BACKGROUND:

The increased risk of hypertension in United States Blacks remains a major unsolved public health problem. Comparisons between macro-population groups in the United States suffer from confounding by social factors and genetic admixture. The study's international comparative design provides a unique opportunity to ascertain the evolution of hypertension among populations with a common genetic background currently living in widely varied social conditions. A well-organized network of investigators currently exists in the societies of the Black diaspora and provides for the first time an opportunity to conduct cross-national research on this question.

DESIGN NARRATIVE:

During the first phase of the project over 12,000 adults between the ages of 25 and 74 were sampled from seven communities: West Africa (Nigeria, urban & rural; Cameroon, urban & rural), the West Indies (St. Lucia, Barbados) and Maywood (lllinois). The screening examination provided information on blood pressure (BP), height, weight, waist/hip ratio, alcohol use, education/occupation, sodium/potassium excretion and social stress. These data provided estimates of hypertension prevalence in each geographic region and the contribution of the known risk factor to higher rates among United States Blacks. In the first phase considerable effort was directed toward establishing a strong research infrastructure in each of the sites and demonstrating the feasibility of cross-national blood pressure comparisons.

In the second phase the research was continued and extended in three areas: 1) Population studies on risk factors. At the start of the study in 1991, it was not clear that adequate procedures were available to allow standardization of mean blood pressure across sites, especially since differences between some sites might be as little as 2 mmHg. Experience since that time suggested that it would be feasible to collect definitive data on this question. In-depth studies were carried out at one of the African sites to investigate the earliest stages of hypertension risk for a population. Investigators in Jamaica and the United Kingdom joined the collaborative group to examine the effect of migration from the Caribbean to the United Kingdom. 2) Prospective study of blood pressure and mortality. It was well known that hypertension accounted for much of the excess mortality among United States Blacks. It was less well recognized, however, that death rates among Blacks in the United States were higher than reported in the Caribbean or Africa. Hypertension was likely to account for that differential. A follow-up study in each region estimated the relative and attributable risk from hypertension. 3) Heredity/Genetics. The populations in this study shared a common ancestral origin in West Africa. Family studies were undertaken to determine the heritability of blood pressure/hypertension within and between sites. In addition, pilot studies on genetic distance and candidate genes for hypertension were conducted.

The study was renewed in FY 1999 to examine in further detail the role of the two most potent hypertensive risk factors, namely dietary sodium and obesity. Randomized studies will be carried out in Nigeria, Jamaica, and Chicago to determine the relative sodium sensitivity of these populations and the factors which condition the blood pressure response. The renin-angiotensin system and renal sodium handling will be compared as causal mechanisms. In addition, body composition will be studied in a large sample of each of the three populations to determine the role of body fat versus lean body mass. Insulin and leptin will be examined and physical activity will be measured by stable isotopes to assess the role of a sedentary lifestyle as a contributor to the hypertension risk experienced by the obese. Existing cohorts will be followed to determine hypertension sequelae and to examine changes in blood pressure with age.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cooper — Loyola University

REFERENCES:
- [Background] Rotimi C, Cooper R, Cao G, Sundarum C, McGee D. Familial aggregation of cardiovascular diseases in African-American pedigrees. Genet Epidemiol. 1994;11(5):397-407. doi: 10.1002/gepi.1370110502. PMID 7835686
- [Background] Rotimi C, Morrison L, Cooper R, Oyejide C, Effiong E, Ladipo M, Osotemihen B, Ward R. Angiotensinogen gene in human hypertension. Lack of an association of the 235T allele among African Americans. Hypertension. 1994 Nov;24(5):591-4. doi: 10.1161/01.hyp.24.5.591. PMID 7960018
- [Background] Cooper RS, Rotimi CN, Kaufman JS, Muna WF, Mensah GA. Hypertension treatment and control in sub-Saharan Africa: the epidemiological basis for policy. BMJ. 1998 Feb 21;316(7131):614-7. doi: 10.1136/bmj.316.7131.614. No abstract available. PMID 9518920
- [Background] Luke AH, Rotimi CN, Cooper RS, Long AE, Forrester TE, Wilks R, Bennett FI, Ogunbiyi O, Compton JA, Bowsher RR. Leptin and body composition of Nigerians, Jamaicans, and US blacks. Am J Clin Nutr. 1998 Mar;67(3):391-6. doi: 10.1093/ajcn/67.3.391. PMID 9497181
- [Background] Kaufman JS, Asuzu MC, Rotimi CN, Johnson OO, Owoaje EE, Cooper RS. The absence of adult mortality data for sub-Saharan Africa: a practical solution. Bull World Health Organ. 1997;75(5):389-95. PMID 9447773
- [Background] Kaufman JS, Asuzu MC, Mufunda J, Forrester T, Wilks R, Luke A, Long AE, Cooper RS. Relationship between blood pressure and body mass index in lean populations. Hypertension. 1997 Dec;30(6):1511-6. doi: 10.1161/01.hyp.30.6.1511. PMID 9403575
- [Background] Kaufman JS, Durazo-Arvizu RA, Rotimi CN, McGee DL, Cooper RS. Obesity and hypertension prevalence in populations of African origin. The Investigators of the International Collaborative Study on Hypertension in Blacks. Epidemiology. 1996 Jul;7(4):398-405. doi: 10.1097/00001648-199607000-00010. PMID 8793366
- [Background] Rotimi C, Luke A, Li Z, Compton J, Bowsher R, Cooper R. Heritability of plasma leptin in a population sample of African-American families. Genet Epidemiol. 1997;14(3):255-63. doi: 10.1002/(SICI)1098-2272(1997)14:33.0.CO;2-4. PMID 9181355
- [Background] Rotimi CN, Cooper RS, Marcovina SM, McGee D, Owoaje E, Ladipo M. Serum distribution of lipoprotein(a) in African Americans and Nigerians: potential evidence for a genotype-environmental effect. Genet Epidemiol. 1997;14(2):157-68. doi: 10.1002/(SICI)1098-2272(1997)14:23.0.CO;2-4. PMID 9129961
- [Background] Forrester T, McFarlane-Anderson N, Bennett FI, Wilks R, Cooper R, Rotimi C, Morrison L, Ward R. The angiotensin converting enzyme and blood pressure in Jamaicans. Am J Hypertens. 1997 May;10(5 Pt 1):519-24. doi: 10.1016/s0895-7061(97)00049-6. PMID 9160762
- [Background] Cooper RS, Rotimi CN, Kaufman JS, Owoaje EE, Fraser H, Forrester T, Wilks R, Riste LK, Cruickshank JK. Prevalence of NIDDM among populations of the African diaspora. Diabetes Care. 1997 Mar;20(3):343-8. doi: 10.2337/diacare.20.3.343. PMID 9051385
- [Background] Rotimi C, Cooper R, Ogunbiyi O, Morrison L, Ladipo M, Tewksbury D, Ward R. Hypertension, serum angiotensinogen, and molecular variants of the angiotensinogen gene among Nigerians. Circulation. 1997 May 20;95(10):2348-50. doi: 10.1161/01.cir.95.10.2348. PMID 9170394
- [Background] Luke A, Durazo-Arvizu R, Rotimi C, Prewitt TE, Forrester T, Wilks R, Ogunbiyi OJ, Schoeller DA, McGee D, Cooper RS. Relation between body mass index and body fat in black population samples from Nigeria, Jamaica, and the United States. Am J Epidemiol. 1997 Apr 1;145(7):620-8. doi: 10.1093/oxfordjournals.aje.a009159. PMID 9098179
- [Background] Kaufman JS, Rotimi CN, Brieger WR, Oladokum MA, Kadiri S, Osotimehin BO, Cooper RS. The mortality risk associated with hypertension: preliminary results of a prospective study in rural Nigeria. J Hum Hypertens. 1996 Jul;10(7):461-4. PMID 8880560
- [Background] Rotimi C, Cooper R. Familial resemblance for anthropometric measurements and relative fat distribution among African Americans. Int J Obes Relat Metab Disord. 1995 Dec;19(12):875-80. PMID 8963355
- [Background] Freeman V, Rotimi C, Cooper R. Hypertension prevalence, awareness, treatment, and control among African Americans in the 1990s: estimates from the Maywood Cardiovascular Survey. Am J Prev Med. 1996 May-Jun;12(3):177-85. PMID 8743873
- [Background] Freeman V, Fraser H, Forrester T, Wilks R, Cruickshank J, Rotimi C, Cooper R. A comparative study of hypertension prevalence, awareness, treatment and control rates in St Lucia, Jamaica and Barbados. J Hypertens. 1996 Apr;14(4):495-501. PMID 8761900
- [Background] Forrester T, McFarlane-Anderson N, Bennet F, Wilks R, Puras A, Cooper R, Rotimi C, Durazo R, Tewksbury D, Morrison L. Angiotensinogen and blood pressure among blacks: findings from a community survey in Jamaica. J Hypertens. 1996 Mar;14(3):315-21. doi: 10.1097/00004872-199603000-00007. PMID 8723984
- [Background] Ataman SL, Cooper R, Rotimi C, McGee D, Osotimehin B, Kadiri S, Kingue S, Muna W, Fraser H, Forrester T, Wilks R. Standardization of blood pressure measurement in an international comparative study. J Clin Epidemiol. 1996 Aug;49(8):869-77. doi: 10.1016/0895-4356(96)00111-4. PMID 8699206
- [Background] Kaufman JS, Owoaje EE, James SA, Rotimi CN, Cooper RS. Determinants of hypertension in West Africa: contribution of anthropometric and dietary factors to urban-rural and socioeconomic gradients. Am J Epidemiol. 1996 Jun 15;143(12):1203-18. doi: 10.1093/oxfordjournals.aje.a008708. PMID 8651219
- [Background] Rotimi C, Puras A, Cooper R, McFarlane-Anderson N, Forrester T, Ogunbiyi O, Morrison L, Ward R. Polymorphisms of renin-angiotensin genes among Nigerians, Jamaicans, and African Americans. Hypertension. 1996 Mar;27(3 Pt 2):558-63. doi: 10.1161/01.hyp.27.3.558. PMID 8613203
- [Background] Cooper RS, Cheng HY, Rotimi C. Basal and stimulated platelet calcium and sodium in hypertensive versus normotensive black people. J Hum Hypertens. 1995 Sep;9(9):747-52. PMID 8551489
- [Background] Okosun IS, Forrester TE, Rotimi CN, Osotimehin BO, Muna WF, Cooper RS. Abdominal adiposity in six populations of West African descent: prevalence and population attributable fraction of hypertension. Obes Res. 1999 Sep;7(5):453-62. doi: 10.1002/j.1550-8528.1999.tb00433.x. PMID 10509602
- [Background] Kaufman JS, Owoaje EE, Rotimi CN, Cooper RS. Blood pressure change in Africa: case study from Nigeria. Hum Biol. 1999 Aug;71(4):641-57. PMID 10453105
- [Background] Okosun IS, Cooper RS, Prewitt TE, Rotimi CN. The relation of central adiposity to components of the insulin resistance syndrome in a biracial US population sample. Ethn Dis. 1999 Spring-Summer;9(2):218-29. PMID 10421084
- [Background] Rotimi CN, Cooper RS, Okosun IS, Olatunbosun ST, Bella AF, Wilks R, Bennett F, Cruickshank JK, Forrester TE. Prevalence of diabetes and impaired glucose tolerance in Nigerians, Jamaicans and US blacks. Ethn Dis. 1999 Spring-Summer;9(2):190-200. PMID 10421081
- [Background] Long AE, Prewitt TE, Kaufman JS, Rotimi CN, Cooper RS, McGee DL. Weight-height relationships among eight populations of West African origin: the case against constant BMI standards. Int J Obes Relat Metab Disord. 1998 Sep;22(9):842-6. doi: 10.1038/sj.ijo.0800670. PMID 9756241
- [Background] Colilla S, Rotimi C, Cooper R, Goldberg J, Cox N. Genetic inheritance of body mass index in African-American and African families. Genet Epidemiol. 2000 Apr;18(4):360-76. doi: 10.1002/(SICI)1098-2272(200004)18:43.0.CO;2-H. PMID 10797595
- [Background] Kaufman JS, Tracy JA, Durazo-Arvizu RA, Cooper RS. Lifestyle, education, and prevalence of hypertension in populations of African origin. Results from the International Collaborative Study on Hypertension in Blacks. Ann Epidemiol. 1997 Jan;7(1):22-7. PMID 9034403
- [Background] Rotimi CN, Cooper RS, Ataman SL, Osotimehin B, Kadiri S, Muna W, Kingue S, Fraser H, McGee D. Distribution of anthropometric variables and the prevalence of obesity in populations of west African origin: the International Collaborative Study on Hypertension in Blacks (ICSHIB). Obes Res. 1995 Sep;3 Suppl 2:95s-105s. doi: 10.1002/j.1550-8528.1995.tb00452.x. PMID 8581794
- [Background] Zhu X, McKenzie CA, Forrester T, Nickerson DA, Broeckel U, Schunkert H, Doering A, Jacob HJ, Cooper RS, Rieder MJ. Localization of a small genomic region associated with elevated ACE. Am J Hum Genet. 2000 Nov;67(5):1144-53. doi: 10.1016/S0002-9297(07)62945-0. Epub 2000 Sep 19. PMID 11001581
- [Background] Cooper R, Forrester T, Ogunbiyi O, Muffinda J. Angiotensinogen levels and obesity in four black populations. ICSHIB Investigators. J Hypertens. 1998 May;16(5):571-5. doi: 10.1097/00004872-199816050-00003. PMID 9797167
- [Background] Luke A, Durazo-Arvizu RA, Rotimi CN, Iams H, Schoeller DA, Adeyemo AA, Forrester TE, Wilks R, Cooper RS. Activity energy expenditure and adiposity among black adults in Nigeria and the United States. Am J Clin Nutr. 2002 Jun;75(6):1045-50. doi: 10.1093/ajcn/75.6.1045. PMID 12036811
- [Background] Collins-Schramm HE, Phillips CM, Operario DJ, Lee JS, Weber JL, Hanson RL, Knowler WC, Cooper R, Li H, Seldin MF. Ethnic-difference markers for use in mapping by admixture linkage disequilibrium. Am J Hum Genet. 2002 Mar;70(3):737-50. doi: 10.1086/339368. Epub 2002 Feb 11. PMID 11845411
- [Background] Zhu X, Bouzekri N, Southam L, Cooper RS, Adeyemo A, McKenzie CA, Luke A, Chen G, Elston RC, Ward R. Linkage and association analysis of angiotensin I-converting enzyme (ACE)-gene polymorphisms with ACE concentration and blood pressure. Am J Hum Genet. 2001 May;68(5):1139-48. doi: 10.1086/320104. Epub 2001 Mar 27. PMID 11283791
- [Background] Adeyemo AA, Prewitt TE, Luke A, Omotade OO, Rotimi CN, Brieger WR, Cooper RS. The feasibility of implementing a dietary sodium reduction intervention among free-living normotensive individuals in south west Nigeria. Ethn Dis. 2002 Spring;12(2):207-12. PMID 12019929
- [Background] Adeyemo AA, Omotade OO, Rotimi CN, Luke AH, Tayo BO, Cooper RS. Heritability of blood pressure in Nigerian families. J Hypertens. 2002 May;20(5):859-63. doi: 10.1097/00004872-200205000-00019. PMID 12011645
- [Background] Lowe WL Jr, Rotimi CN, Luke A, Guo X, Zhu X, Comuzzie AG, Schuh TS, Halbach S, Kotlar TJ, Cooper RS. The beta 3-adrenergic receptor gene and obesity in a population sample of African Americans. Int J Obes Relat Metab Disord. 2001 Jan;25(1):54-60. doi: 10.1038/sj.ijo.0801487. PMID 11244458
- [Background] Luke A, Rotimi CN, Adeyemo AA, Durazo-Arvizu RA, Prewitt TE, Moragne-Kayser L, Harders R, Cooper RS. Comparability of resting energy expenditure in Nigerians and U.S. blacks. Obes Res. 2000 Aug;8(5):351-9. doi: 10.1038/oby.2000.42. PMID 10968726
- [Background] Okosun IS, Liao Y, Rotimi CN, Prewitt TE, Cooper RS. Abdominal adiposity and clustering of multiple metabolic syndrome in White, Black and Hispanic americans. Ann Epidemiol. 2000 Jul;10(5):263-70. doi: 10.1016/s1047-2797(00)00045-4. PMID 10942873
- [Background] Schork NJ, Chakravarti A, Thiel B, Fornage M, Jacob HJ, Cai R, Rotimi CN, Cooper RS, Weder AB. Lack of association between a biallelic polymorphism in the adducin gene and blood pressure in whites and African Americans. Am J Hypertens. 2000 Jun;13(6 Pt 1):693-8. doi: 10.1016/s0895-7061(00)00237-5. PMID 10912755
- [Background] Okosun IS, Liao Y, Rotimi CN, Dever GE, Cooper RS. Impact of birth weight on ethnic variations in subcutaneous and central adiposity in American children aged 5-11 years. A study from the Third National Health and Nutrition Examination Survey. Int J Obes Relat Metab Disord. 2000 Apr;24(4):479-84. doi: 10.1038/sj.ijo.0801182. PMID 10805505
- [Background] Okosun IS, Liao Y, Rotimi CN, Choi S, Cooper RS. Predictive values of waist circumference for dyslipidemia, type 2 diabetes and hypertension in overweight White, Black, and Hispanic American adults. J Clin Epidemiol. 2000 Apr;53(4):401-8. doi: 10.1016/s0895-4356(99)00217-6. PMID 10785571
- [Background] Collins-Schramm HE, Kittles RA, Operario DJ, Weber JL, Criswell LA, Cooper RS, Seldin MF. Markers that discriminate between European and African ancestry show limited variation within Africa. Hum Genet. 2002 Dec;111(6):566-9. doi: 10.1007/s00439-002-0818-z. Epub 2002 Sep 14. PMID 12436248
- [Background] Cooper RS, Luke A, Zhu X, Kan D, Adeyemo A, Rotimi C, Bouzekri N, Ward R. Genome scan among Nigerians linking blood pressure to chromosomes 2, 3, and 19. Hypertension. 2002 Nov;40(5):629-33. doi: 10.1161/01.hyp.0000035708.02789.39. PMID 12411454
- [Background] Cox R, Bouzekri N, Martin S, Southam L, Hugill A, Golamaully M, Cooper R, Adeyemo A, Soubrier F, Ward R, Lathrop GM, Matsuda F, Farrall M. Angiotensin-1-converting enzyme (ACE) plasma concentration is influenced by multiple ACE-linked quantitative trait nucleotides. Hum Mol Genet. 2002 Nov 1;11(23):2969-77. doi: 10.1093/hmg/11.23.2969. PMID 12393808
- [Background] Sargeant LA, Bennett FI, Forrester TE, Cooper RS, Wilks RJ. Predicting incident diabetes in Jamaica: the role of anthropometry. Obes Res. 2002 Aug;10(8):792-8. doi: 10.1038/oby.2002.107. PMID 12181388
- [Background] Leman CR, Adeyemo AA, Schoeller DA, Cooper RS, Luke A. Body composition of children in south-western Nigeria: validation of bio-electrical impedance analysis. Ann Trop Paediatr. 2003 Mar;23(1):61-7. doi: 10.1179/000349803125002887. PMID 12648327
- [Background] Adeyemo A, Luke A, Cooper R, Wu X, Tayo B, Zhu X, Rotimi C, Bouzekri N, Ward R. A genome-wide scan for body mass index among Nigerian families. Obes Res. 2003 Feb;11(2):266-73. doi: 10.1038/oby.2003.40. PMID 12582223
- [Background] Zhu X, Cooper RS. Linkage disequilibrium analysis of the renin-angiotensin system genes. Curr Hypertens Rep. 2003 Feb;5(1):40-6. doi: 10.1007/s11906-003-0009-x. PMID 12530934
- [Background] Mendez MA, Cooper R, Wilks R, Luke A, Forrester T. Income, education, and blood pressure in adults in Jamaica, a middle-income developing country. Int J Epidemiol. 2003 Jun;32(3):400-8. doi: 10.1093/ije/dyg083. PMID 12777427
- [Background] Luke A, Wu X, Zhu X, Kan D, Su Y, Cooper R. Linkage for BMI at 3q27 region confirmed in an African-American population. Diabetes. 2003 May;52(5):1284-7. doi: 10.2337/diabetes.52.5.1284. PMID 12716766
- [Background] Thiel BA, Chakravarti A, Cooper RS, Luke A, Lewis S, Lynn A, Tiwari H, Schork NJ, Weder AB. A genome-wide linkage analysis investigating the determinants of blood pressure in whites and African Americans. Am J Hypertens. 2003 Feb;16(2):151-3. doi: 10.1016/s0895-7061(02)03246-6. PMID 12559684
- [Background] Cooper RS. Gene-environment interactions and the etiology of common complex disease. Ann Intern Med. 2003 Sep 2;139(5 Pt 2):437-40. doi: 10.7326/0003-4819-139-5_part_2-200309021-00011. PMID 12965972
- [Background] Boyne MS, Sargeant LA, Bennett FI, Cooper RS, Wilks RJ, Forrester TE. Features of isolated post-challenge hyperglycaemia in Jamaican adults. West Indian Med J. 2004 Jan;53(1):7-11. PMID 15114886
- [Background] Bouzekri N, Zhu X, Jiang Y, McKenzie CA, Luke A, Forrester T, Adeyemo A, Kan D, Farrall M, Anderson S, Cooper RS, Ward R. Angiotensin I-converting enzyme polymorphisms, ACE level and blood pressure among Nigerians, Jamaicans and African-Americans. Eur J Hum Genet. 2004 Jun;12(6):460-8. doi: 10.1038/sj.ejhg.5201166. PMID 14970846
- [Background] Lawoyin TO, Asuzu MC, Kaufman J, Rotimi C, Johnson L, Owoaje E, Cooper R. Using verbal autopsy to identify and proportionally assign cause of death in Ibadan, southwest Nigeria. Niger Postgrad Med J. 2004 Sep;11(3):182-6. PMID 15505646
- [Background] Sargeant LA, Boyne MS, Bennett FI, Forrester TE, Cooper RS, Wilks RJ. Impaired glucose regulation in adults in Jamaica: who should have the oral glucose tolerance test? Rev Panam Salud Publica. 2004 Jul;16(1):35-42. doi: 10.1590/s1020-49892004000700005. PMID 15333264
- [Background] Koivukoski L, Fisher SA, Kanninen T, Lewis CM, von Wowern F, Hunt S, Kardia SL, Levy D, Perola M, Rankinen T, Rao DC, Rice T, Thiel BA, Melander O. Meta-analysis of genome-wide scans for hypertension and blood pressure in Caucasians shows evidence of susceptibility regions on chromosomes 2 and 3. Hum Mol Genet. 2004 Oct 1;13(19):2325-32. doi: 10.1093/hmg/ddh237. Epub 2004 Aug 4. PMID 15294874
- [Background] Fejerman L, Bouzekri N, Wu X, Adeyemo A, Luke A, Zhu X, Ward R, Cooper RS. Association between evolutionary history of angiotensinogen haplotypes and plasma levels. Hum Genet. 2004 Sep;115(4):310-8. doi: 10.1007/s00439-004-1141-7. PMID 15278435
- [Background] Boyne MS, Gaskin P, Luke A, Wilks RJ, Bennett FI, Younger N, Sargeant LA, Adeyemo AA, Cooper RS, Forrester TE. Energetic determinants of glucose tolerance status in Jamaican adults. Eur J Clin Nutr. 2004 Dec;58(12):1666-8. doi: 10.1038/sj.ejcn.1602011. PMID 15162140
- [Background] Mendez MA, Wynter S, Wilks R, Forrester T. Under- and overreporting of energy is related to obesity, lifestyle factors and food group intakes in Jamaican adults. Public Health Nutr. 2004 Feb;7(1):9-19. doi: 10.1079/phn2003508. PMID 14972067
- [Background] Mendez MA, Cooper RS, Luke A, Wilks R, Bennett F, Forrester T. Higher income is more strongly associated with obesity than with obesity-related metabolic disorders in Jamaican adults. Int J Obes Relat Metab Disord. 2004 Apr;28(4):543-50. doi: 10.1038/sj.ijo.0802584. PMID 14770191
- [Background] Luke A, Adeyemo A, Kramer H, Forrester T, Cooper RS. Association between blood pressure and resting energy expenditure independent of body size. Hypertension. 2004 Mar;43(3):555-60. doi: 10.1161/01.HYP.0000118020.44335.20. Epub 2004 Feb 2. PMID 14757780
- [Background] McKenzie CA, Sinsheimer JS, Adeyemo AA, Cox RD, Southam L, Hugill A, Bouzekri N, Lathrop M, Forrester TE, Cooper RS, Ward R. SNP haplotypes in the angiotensin I-converting enzyme (ACE) gene: analysis of Nigerian family data using gamete competition models. Ann Hum Genet. 2005 Mar;69(Pt 2):227-32. doi: 10.1046/j.1529-8817.2004.00142.x. PMID 15720304
- [Background] Zhu X, Fejerman L, Luke A, Adeyemo A, Cooper RS. Haplotypes produced from rare variants in the promoter and coding regions of angiotensinogen contribute to variation in angiotensinogen levels. Hum Mol Genet. 2005 Mar 1;14(5):639-43. doi: 10.1093/hmg/ddi060. Epub 2005 Jan 13. PMID 15649942
- [Background] Cooper R, Rotimi C. Hypertension in blacks. Am J Hypertens. 1997 Jul;10(7 Pt 1):804-12. doi: 10.1016/s0895-7061(97)00211-2. PMID 9234837